CLINICAL TRIAL: NCT02104336
Title: An Open-Label Phase 2 Safety and Efficacy Study of EPI-743 (VincerinoneTM) in Children With Pearson Syndrome
Brief Title: Phase 2 Study of EPI-743 in Children With Pearson Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Results from other studies did not support continuation of this trial
Sponsor: Edison Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPI743-13-024
Record Dates: First submitted 2014-04-02; First posted 2014-04-04 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Pearson Syndrome
Keywords: Pearson; EPI743; EPI-743; Vincerinone; Mitochondrial disorder; Mitochondrial disease
MeSH Terms: conditions — VLCAD deficiency; Mitochondrial Diseases | interventions — alpha-tocotrienol quinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EPI-743 (Experimental): 15 mg/kg EPI-743 to be administered three times per day for 1 year
  Interventions: Drug: EPI-743

INTERVENTIONS:
Drug: EPI-743 — EPI-743 is the quinone oxidation product of alpha-tocotrienol
  Other Names: Vincerinone (TM)

SUMMARY:
Treatment of Pediatric Subjects with Pearson syndrome

DETAILED DESCRIPTION:
If effective, treatment with EPI-743 should result in a significant reduction in occurrence of sepsis, metabolic crisis, hepatic failure and transfusion dependence.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed diagnosis of Pearson syndrome
* Age less than 18
* Availability of medical history for 12 months prior to enrollment
* Abstention from use of CoQ10, vitamin E, lipoic acid and Idebenone 14 days prior to treatment with EPI-743

Exclusion Criteria:

* Allergy to EPI-743, sesame oil or vitamin E
* Clinical history of bleeding/ abnormal PT/PTT
* Concurrent inborn errors of metabolism
* Use of anticoagulant medications
* Participation in any interventional study within 30 days of treatment
* Use of erythropoietin 30 days prior to trial enrollment

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2014-08-31 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2016-02-29 (Actual)

PRIMARY OUTCOMES:
Occurence of episodes of sepsis, metabolic crisis or hepatic faillure | 1 year

SECONDARY OUTCOMES:
Transfusion avoidance | 1 year
Hematologic function | 1 year
Neuromuscular function | 1 year
  Neuromuscular function as assessed by Gross Motor Function Measure
Disease severity | 1 year
  Disease severity as assessed by Newcastle Pediatric Mitochondrial Disease Scale
Renal function | 1 year
Hepatic function | 1 year
Weight gain | 1 year
Hospitalizations | 1 year
Pancreatic function | 1 year
  Pancreatic function as assessed by insulin requirement and hemoglobin A1c
Mortality | 1 year

OTHER OUTCOMES:
Number of Dose Limiting SAEs | 1 year
  Any adverse event greater than or equal to grade 3 that is deemed related to treatment with EPI-743 and not related to underlying disease

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Klein, MD, FACS, Study Chair — Edison Pharmaceuticals
Locations (4):
- United States (4):
  - Children's Hospital of Orange County, Orange, California
  - Cleveland Clinic, Cleveland, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas